CLINICAL TRIAL: NCT00000265
Title: Subjective Effects of Nitrous Oxide in Dental Patients
Brief Title: Subjective Effects of Nitrous Oxide in Dental Patients - 17
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: NIDA-08391-17; R01DA008391 (NIH); R01-08391-17
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; anxiety; subjective effects; dental; patients
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Low anxiety
- Moderate anxiety
- High anxiety

SUMMARY:
The purpose of this study was to characterize mood changes during nitrous oxide inhalation in patients with different levels of preoperative dental anxiety.

ELIGIBILITY:
Please contact site for information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1997-07; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Anxiety scale | Before, during, after dental procedure
Mood scale | Before, during, after dental procedure

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States